CLINICAL TRIAL: NCT00742365
Title: Predicting Light Treatment's Effectiveness on Reducing Depression and Cardiovascular Risk in Seasonal Affective Disorder
Brief Title: Predicting Effectiveness of Light Treatment for Winter Seasonal Affective Disorder
Status: Completed | Type: Observational
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Teodor Postolache, Principal Investigator, University of Maryland, Baltimore
Other Study IDs: HP-00043574; R34MH073797 (NIH); DSIR 83-ATSO; H-28845
Record Dates: First submitted 2008-08-25; First posted 2008-08-27 (Estimated); Last update posted 2019-11-21 (Actual); Status verified 2019-11

CONDITIONS: Depression
Keywords: Seasonal Affective Disorder; Light Therapy; Seasonal Depression; Psychiatric Disorder; Bright Light; Major Depressive Disorder; Bipolar Disorder
MeSH Terms: conditions — Depression; Seasonal Affective Disorder; Mental Disorders; Depressive Disorder, Major; Bipolar Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- A: Participants will be given a 1-hour lab test of bright light treatment, then the bright light treatment for 6 weeks.
  Interventions: Device: Bright light
- B: Participants will be given a 1-hour treatment of the red light placebo, then the bright light treatment for 6 weeks.
  Interventions: Device: Red light placebo

INTERVENTIONS:
Device: Bright light — One hour of exposure to bright light daily upon awakening for 6 weeks.
  Other Names: Brite light III light box (Apollo) 10,000 lux.
  Groups: A
Device: Red light placebo — One hour of exposure to red light.
  Other Names: Dim red light box (Apollo) 50 lux.
  Groups: B

SUMMARY:
This study will evaluate a possible tool for predicting future effectiveness of bright light in treating seasonal affective disorder, winter subtype, and will examine secondary effects of bright light on cardiovascular risk factors.

DETAILED DESCRIPTION:
The winter subtype of seasonal affective disorder (SAD) is characterized by episodes of major depression in the fall and winter, with remission of these episodes in the spring and summer. SAD disrupts the lives of millions of Americans, who experience symptoms such as restless agitation, increased appetite and weight gain, and reduced energy and motivation. Bright light treatment, while shown to be effective in improving SAD in 75% of cases, only causes a full remission in 50% of cases. If doctors had a diagnostic tool to determine which patients would respond to bright light therapy, they could make better decisions about whether to prescribe bright light as treatment. This study will examine a possible diagnostic tool-a single, 1-hour bright light session-for predicting improvement in SAD symptoms over an extended course of bright light treatment. Additionally, because many symptoms of SAD (like weight gain and sedentary lifestyle) correspond to cardiovascular risk, this study will examine whether bright light treatment correlates with improved cardiovascular health.

Participants with SAD will be randomly assigned to first receive a 1-hour session of either bright light or the placebo, red light. Then all participants will switch and receive a 1-hour session of the other type of light. Red light has been accepted as a placebo in previous SAD studies because it does not suppress melatonin or shift circadian rhythms. Before and after each light session, participants will have their SAD symptoms evaluated in a clinical interview and self-report measure. After these two light sessions, all participants will receive instructions for administering bright light treatment on their own at home. For the next 6 weeks, participants will administer the bright light to themselves for 1 hour every morning. Every week they will undergo clinical interviews by phone and will mail in self-report measures, some completed daily and some weekly, to the researchers. The participants will have checkups and interviews in person on Weeks 4 and 6. At the two time periods, SAD symptoms and indicators of cardiovascular risk, such as appetite and sleep loss, will be evaluated. The participant responses to bright light and red light at the initial session will be compared with the participant responses to the subsequent 6-week treatment.

ELIGIBILITY:
Inclusion Criteria:

* Current major depressive disorder, by structured diagnostic interview (SCID), or current bipolar II disorder, if no prior history of rapid cycling, by SCID
* Prior history of major depressive disorder or bipolar II disorder with seasonal specifier, by SCID
* Score of 21 or greater on Hamilton Rating Scale for Depression - Seasonal Affective Disorder Version (SIGH-SAD), met at three time points (informed consent session, 24 hours prior to first light therapy session, and at first light therapy session)

Exclusion Criteria:

* Current bipolar I disorder, psychotic disorder, or cognitive disorder, by SCID
* Illicit drug use in the past year, by self-report, or alcohol abuse by SCID
* History of systemic lupus erythematosus
* History of heart attack or stroke
* No antidepressant, mood stabilizer, or antipsychotic medication treatment 30 days before treatment
* Current occupation involves shift work
* Current sensitivity to bright light or vision problems not correctable by glasses, by self-report
* Inability to distinguish colors or see stars at night because of increased light sensitivity, by self-report
* Current suicidal ideation, by self-report during SCID interview
* Women of childbearing potential who are pregnant, nursing, or trying to become pregnant. Female participants of childbearing potential must agree to one of the following types of birth control: oral, transdermal, or implantable hormonal contraceptives; intrauterine device; diaphragm plus spermicide; or female condom plus spermicide.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with history of recurrent winter depression
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2007-11; Primary Completion 2010-04 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Hamilton rating scale for depressional seasonal affective disorder (SIGH SAD) | Measured at baseline, 1 hour after light treatment, and weekly for 6 weeks

SECONDARY OUTCOMES:
Hunger questionnaire | Measured daily for 6 weeks
Three factor eating questionnaire | Measured weekly for 6 weeks
Sleep log | Measured weekly for 6 weeks
Food craving questionnaire | Measured daily for 6 weeks
Side effects questionnaire | Measured weekly for 6 weeks
Adherence questionnaire | Measured weekly for 6 weeks
Profile of Mood States | Measured at baseline, 1 hour after light treatment, and weekly for 6 weeks
Beck Depression Inventory-II (BDI) | Measured at baseline, 1 hour after light treatment, and weekly for 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Teodor T. Postolache, MD, Principal Investigator — University of Maryland, Baltimore

REFERENCES:
- [Background] Uzoma HN, Reeves GM, Langenberg P, Khabazghazvini B, Balis TG, Johnson MA, Sleemi A, Scrandis DA, Zimmerman SA, Vaswani D, Nijjar GV, Cabassa J, Lapidus M, Rohan KJ, Postolache TT. Light treatment for seasonal Winter depression in African-American vs Caucasian outpatients. World J Psychiatry. 2015 Mar 22;5(1):138-46. doi: 10.5498/wjp.v5.i1.138. PMID 25815263
- [Background] Reeves GM, Rohan KJ, Langenberg P, Snitker S, Postolache TT. Calibration of response and remission cut-points on the Beck Depression Inventory-Second Edition for monitoring seasonal affective disorder treatment outcomes. J Affect Disord. 2012 Apr;138(1-2):123-7. doi: 10.1016/j.jad.2011.12.003. Epub 2012 Jan 25. PMID 22277151
- [Background] Reeves GM, Nijjar GV, Langenberg P, Johnson MA, Khabazghazvini B, Sleemi A, Vaswani D, Lapidus M, Manalai P, Tariq M, Acharya M, Cabassa J, Snitker S, Postolache TT. Improvement in depression scores after 1 hour of light therapy treatment in patients with seasonal affective disorder. J Nerv Ment Dis. 2012 Jan;200(1):51-5. doi: 10.1097/NMD.0b013e31823e56ca. PMID 22210362
- [Background] Virk G, Reeves G, Rosenthal NE, Sher L, Postolache TT. Short exposure to light treatment improves depression scores in patients with seasonal affective disorder: A brief report. Int J Disabil Hum Dev. 2009 Jul;8(3):283-286. doi: 10.1901/jaba.2009.8-283. PMID 20686638